CLINICAL TRIAL: NCT06843928
Title: The Adjunctive Effect of a Titanium Brush in the Non-Surgical Treatment of Peri-Implantitis: a Randomized Multi-Center Controlled Clinical Trial
Brief Title: The Adjunctive Effect of a Titanium Brush in the Non-Surgical Treatment of Peri-Implantitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Javi Vilarrasa, Clinical Professor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PER-ECL-2024-05
Record Dates: First submitted 2024-12-18; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-12

CONDITIONS: Peri-implantitis; Titanium Brush; Non-surgical Submucosal Debridement
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Participants will receive submucosal debridement alone
  Interventions: Device: Submucosal debridement; Device: Submucosal debridement + titanium brushes
- Test Group (Experimental): Participants will receive submucosal debridement and titanium brushes
  Interventions: Device: Submucosal debridement; Device: Submucosal debridement + titanium brushes

INTERVENTIONS:
Device: Submucosal debridement — Participants will undergo non-surgical submucosal debridement alone (SD)
Device: Submucosal debridement + titanium brushes — Participants will undergo non-surgical submucosal debridement + titanium brushes (SD+TiBr)

SUMMARY:
Peri-implantitis is a plaque-associated condition occurring around dental implants, characterized by inflammation in the peri-implant mucosa and loss of supporting bone. To stop this progression, mechanical debridement of biofilm and calculus is commonly used to treat peri-implant lesions as well as the use of adjunctive measures such as titanium brushes. As observed, they improved plaque removal when compared with steel curettes alone. Therefore, it is of interest to evaluate the impact of this procedure in terms of clinical, radiographic and microbiological outcomes to assess their efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with ≥18 years of age.
* Ability to understand all the study procedures and to comply with them along the entire study period. Ability and willingness to give written informed consent.
* An adequate level of oral hygiene (plaque index ≤ 25%) (O'Leary et al., 1972).
* Treated periodontal disease.
* Presence of at least one titanium implant with peri-implantitis [i.e., presence of bleeding and/or suppuration on gentle probing with probing depth of ≥6 mm, and progressive bone loss. In the absence of initial radiographs, a bone level ≥2 mm apical to the most coronal part of the intrabony portion of the implant will be used as threshold of disease (Romandini et al., 2021)].
* Horizontal and vertical peri-implant bone defects.
* Implant function time ≥ 1 year.
* Presence of ≥2mm of keratinized peri-implant mucosa.
* Screw-retained single and multiple restorations.

Exclusion Criteria:

* Untreated periodontitis.
* Smokers > 10 cigarettes per day.
* Local or systemic diseases that would interfere with routine periodontal therapy (i.e., uncontrolled diabetes mellitus, cancer, HIV, chronic high-dose steroid therapy, metabolic bone disease, radiation, immunosuppressive disease, hepatic dysfunction, immunosuppressive disease, autoimmune disease).
* Pregnant or lactating women.
* Previous surgical and non-surgical treatment of affected implants at least 12 months prior to the beginning of the study.
* Radiographic peri-implant bone loss > two-thirds.
* Mobility of the implant.
* Known allergy or intolerance to macrolides.
* Use of systemic antibiotics during the last 3 months.
* Need of endocarditis prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-07-17 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Pocket depth changes | 12 Months
  The primary outcome variable will be pocket depth changes at 1 year of follow-up.

SECONDARY OUTCOMES:
Full mouth plaque index (FMPI) | 12 Months
  Assessed dichotomously as presence or absence of plaque will be scored if present along the gingival margin and if it can be removed with the side of the probe. The percentage of surfaces with plaque out of the total number of examined tooth surfaces will be calculated.
Full mouth bleeding index (FMBI) | 12 Months
  Assessed dichotomously as presence or absence of bleeding after 30 seconds of gently probing. The proportion of bleeding surfaces out of the total number of examined surfaces will be calculated.
Modified plaque index (mPI) | 12 Months
  * Score 0: no detection of plaque.
  * Score 1: plaque only recognized by running a probe across the smooth marginal surface of the implant.
  * Score 2: plaque can be seen by the naked eye.
  * Score 3: abundance of soft matter.
Modified bleeding index (mBI) | 12 Months
  * Score 0: no bleeding.
  * Score 1: isolated bleeding spots visible.
  * Score 2: blood forms a confluent red line on margin.
  * Score 3: heavy or profuse bleeding.
Suppuration on probing (SoP) | 12 Months
  Presence or absence of suppuration after gentle probing.
Mucosal recession (MR) | 12 Months
  Distance (mm) from the mucosal margin and the interface between implant and abutment.
Keratinized mucosa (KM) | 12 Months
  Distance (mm) from the mucosal margin to the mucogingival junction at the midbuccal aspect of the implant.
Radiographic parameters | 12 Months
  Marginal bone level (MBL): distance (mm) between the implant shoulder and the base of the defect at the mesial and distal aspect.
Radiographic parameters | 12 Months
  Intra-bony defect (ID): distance (mm) between the bottom of the defect and the line connecting the distal and mesial inter-proximal bone crest.
Radiographic parameters | 12 Months
  Intra-bony defect width (WD): distance (mm) between the distal and mesial inter- proximal bone crest and the implant surface.
Radiographic parameters | 12 Months
  Angulation of the intra-bony defect (AD): angle resulted from a vertical line along the outer implant surface and a line extending along the peri-implant bone defect.
Microbiological analysis | 12 Months
  Total bacterial load (CFU/ml) Microbiome alpha-diversity
Microbiological analysis | 12 Months
  Total bacterial load (CFU/ml) Microbiome beta-diversity
Microbiological analysis | 12 Months
  Total bacterial load (CFU/ml) Relative and differential bacterial genera abundance at different timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No